CLINICAL TRIAL: NCT04654962
Title: Use of Anesthetic Block for the Prevention of in Hospital Delirium in Patients of the Orthogeriatric Clinical Care Center of the Fundacion Santa fe de Bogotá University Hospital and Infantil San Jose University Hospital From 2019 - 2020
Brief Title: Use of Anesthetic Block for the Prevention of in Hospital Delirium in Patients of the Orthogeriatric Clinical Care Center of the HUFSFB and HUSJI From 2019 - 2020
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Jonathan Tihanyi Feldman, Clinical research assistant of the Orthogeriatric Clinical Care Center, Fundación Santa Fe de Bogota
Other Study IDs: CEIS-2020-083
Record Dates: First submitted 2020-11-25; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Delirium in Old Age; Fragility Fracture; Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients receiving preoperative analgesic management with anesthetic block: This cohort includes all patients that received preoperative anesthetic block for hip fracture surgery as main analgesic management during the study period.
  Interventions: Procedure: Anesthetic nerve block
- patients receiving conventional preoperative analgesic management: This cohort includes all patients that received conventional preoperative analgesic management (oral, intravenous or intramuscular medication) for hip fracture surgery as main analgesic management during the study period.

INTERVENTIONS:
Procedure: Anesthetic nerve block — iliac fascia block is an analgesic technique that uses local anesthesia, is effective and relatively safe in preoperative management. The target of this block is the femoral and lateral femoral cutaneous nerves; which innervate the anterior aspect of the thigh, as well as the muscle and periosteum that covers the femoral head, neck and proximal femur.
  Groups: patients receiving preoperative analgesic management with anesthetic block

SUMMARY:
The purpose of this study is to identify the association between analgesic management with blockade of the iliac fascia versus intravenous analgesia with the presence of delirium during hospital stay in patients admitted to the orthogeriatric clinical care center, to determine the opioid consumption of both groups of patients during hospitalization and determine the risk factors that may be associated with a greater presentation of delirium.

DETAILED DESCRIPTION:
Nowadays, with the increase in the geriatric population, there is evidence of an increase in the prevalent conditions in this group, finding within them fragility hip fractures. Additionally, most of these patients have a large number of associated comorbidities, which may require greater specialization in care.

To reduce the possible complications that may be related, different management protocols have been implemented, including pain management strategies such as preventive analgesics, regional blocks, and early surgery. Conventional treatment with the use of intravenous medications can have unwanted effects in geriatric patients with hip fracture, especially in those with greater comorbidity, since medications such as opioids can cause multiple adverse effects, including delirium. Also, not treating pain properly can cause complications such as depression and ulcers in addition to delirium.

This is why the objective of this study is to define whether there is any association between the presentation of delirium in patients over 65 years of age with hip fracture who undergo iliac fascia block upon admission compared to those who receive only IV analgesia Therefore, this retrospective cohort study will be carried out with which it is sought to contribute to the knowledge to continue carrying out early pain management, with the aim of achieving better pain control, a decrease in opioid consumption and thus having a lower number of patients with delirium during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age with a diagnosis of hip fracture due to fragility who are admitted to the Orthogeriatric clinical care center at the Santa Fe de Bogotá Foundation and the San José Infantil University Hospital between January 2019 and December 2020. These two institutions are selected Since they have a model of care for this type of patient, it is similar and therefore comparable.

Exclusion Criteria:

* Patients diagnosed with delirium on admission to the emergency room.
* Patients with hip fracture caused by high energy trauma
* Patients with hip fracture related with tumoral disease or metastasis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: * Patients older than 65 years with a diagnosis of hip fracture who are admitted to the Orthogeriatric Clinical Care Center at the Santa Fe de Bogotá Foundation in a period between January 2019 and December 2020.
  * Patients over 65 years of age with a diagnosis of hip fracture who enter the Excellence Program in Orthogeriatrics at the San José Infantil University Hospital in a period between January 2019 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
In hospital Delirium | Through study completion, an average of 1 year
  Presence of delirium measured with the Confusion Assessment Method (CAM) scale during hospitalization. The CAM scale assesses the presence and severity of delirium, and its algorithm is based on four main features of delirium: 1) acute onset and fluctuating course, 2) inattention, 3) disorganized thinking, and 4) altered level of consciousness. A diagnosis of delirium according to the CAM requires the presence of features 1, 2, and either 3 or 4.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Olarte, MD, Principal Investigator — Orthopedic surgeon
Locations (1):
- Hospital Universitario Fundación Santa fe de Bogotá, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided